CLINICAL TRIAL: NCT04407520
Title: Survival of Direct Composite Restorations Placed Under General Anesthesia in Adult Patients With Intellectual and/or Physical Disabilities and Risk Factors for Repeated Dental Treatment in General Anesthesia of Adult Patients With Intellectual and/or Physical Disabilities
Brief Title: Retrospective Database Study: Survival of Direct Composite Restorations Placed Under General Anesthesia in Adult Patients With Intellectual and/or Physical Disabilities and Risk Factors for Repeated Dental Treatment in General Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, PD Dr. med. dent., Dr. rer. medic., Senior Dental Practitioner, University Medical Center Goettingen
Other Study IDs: Survival-Disabled; 15/1/18 (Other: Local Ethics Commission)
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Intellectual and/or Physical Disabilities; Dental Treatment Under General Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with intellectual and/or physical disabilities: Adult patients with intellectual and/or physical disabilities requiring dental treatment under general anesthesia
  Interventions: Other: No patient treatment is associated with the study

INTERVENTIONS:
Other: No patient treatment is associated with the study — No patient treatment is associated with the study.

SUMMARY:
The aim of this study is to assess the survival of direct anterior and/or posterior composite restoration placed in general anesthesia in permanent teeth of adult patients with intellectual and/or physical disabilities. Further aim is to identify potential risk factors predicting repeated dental treatment under general anesthesia.

Survival of composite restorations placed under general anesthesia in adult patients with intellectual and/or physical disabilities between 2011 and 2019 will be retrospectively analysed. Failure is defined as the need for replacement of at least one surface of the original restoration or extraction of the tooth. Individual-, tooth- and restoration-related factors are obtained from digital and paper-based dental records. Mean annual failure rates (mAFR) and median survival time will be calculated (Kaplan-Meier statistics). The effect of potential risk factors on failure will be tested using univariate log-rank tests and multivariate Cox-regression analysis.

Adult patients with intellectual and/or physical disabilities who received dental treatment under general anesthesia between 2011 and 2017 will be retrospectively analyzed. Demographic, anamnestic, oral health and treatment factors will be obtained from digital and paper-based dental records. Duration of intervals without a subsequent dental treatment under general anesthesia will be assessed using Kaplan-Meier statistics. Potential predictive factors will be tested using log-rank tests and multi-variate Cox-regression analysis.

DETAILED DESCRIPTION:
No patient treatment is associated with the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with intellectual and/or physical disabilities that were treated under general anesthesia in the Department of Preventive Dentistry, Periodontology and Cariology between January 2011 and December 2019

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with intellectual and/or physical disabilities and need for dental treatment under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2011-01-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Failure of restoration placed under general anesthesia | 2011-2019
  Failure is defined as the need for replacement of at least one surface of the original restoration or extraction of the tooth.

SECONDARY OUTCOMES:
Repeated dental treatment under general anesthesia | 2011-2017

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maes MS, Kanzow P, Hrasky V, Wiegand A. Survival of direct composite restorations placed under general anesthesia in adult patients with intellectual and/or physical disabilities. Clin Oral Investig. 2021 Jul;25(7):4563-4569. doi: 10.1007/s00784-020-03770-y. Epub 2021 Jan 15. PMID 33449193
- [Result] Maes MS, Kanzow P, Biermann J, Leha A, Hrasky V, Wiegand A. Risk factors for repeated general anesthesia for dental treatment of adult patients with intellectual and/or physical disabilities. Clin Oral Investig. 2022 Feb;26(2):1695-1700. doi: 10.1007/s00784-021-04142-w. Epub 2021 Aug 25. PMID 34432139